CLINICAL TRIAL: NCT06716164
Title: Safety and Efficacy of Metabolically Armed CD19 CAR-T Cells (Meta10-19) in the Treatment of r/r B-NHL Clinical Research
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Meta10-19-006
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: Meta10-19; CAR-T Cells Therapy; B-cell Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Metabolically Armed CD19 CAR-T cells (Experimental): Patients or donors undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CAR-T cells infusion. A dose of metabolically armed CD19 CAR-T cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed CD19 CAR-T cells

INTERVENTIONS:
Drug: Metabolically Armed CD19 CAR-T cells — Each subject receive metabolically armed CD19 CAR- T cells by intravenous infusion.
  Other Names: Meta10-19

SUMMARY:
A Study of Metabolically Armed CD19 CAR-T Cells Therapy for Patients With Relapsed and/or Refractory B-cell Non-Hodgkin lymphoma

DETAILED DESCRIPTION:
This is a single arm,open-label study.This study is indicated for relapsed and/or refractory B-cell Non-Hodgkin lymphoma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products and our earlier disclosed clinical trials.

1. Main research objectives:

   To evaluate the safety and efficacy of metabolically armed CD19 CAR-T Cells in the treatment of r/r B-NHL.
2. Secondary research objectives:

   * To evaluate the pharmacokinetic (PK) and pharmacodynamics(PD) characteristics of metabolically armed CD19 CAR-T Cells after infusion.
   * To evaluate tumor remission after infusion of metabolically armed CD19 CAR-T Cells.

ELIGIBILITY:
Inclusion Criteria:

* All subjects or guardians must sign an informed consent form approved by the Ethics Committee in person before commencing any screening process;
* Age > 18 years old, ≤ 70 years old, male or female;
* Diagnosis of relapsed/refractory (R/R) indolent B-cell lymphoma, and/or R/R diffuse large B-cell lymphoma (DLBCL). Refractory diseases are defined as one of the following：

  1. Patients with relapsed or refractory B-cell lymphoma treated with one standard treatment regimen and one salvage regimen treated with rituximab or another CD20 antibody drug and at least two treatment regiments appropriate for their disease, one of which should include anthracyclines;
  2. After treatment with these regimens, patients maintain SD (SD duration ≤ 12 months) or still progress；
  3. Recurrence after autologous hematopoietic stem cell transplantation, or recurrence of allogeneic HSCT, or inability to accept HSCT for various reasons；
  4. Patients with double-strike or triple-strike B-cell lymphoma who did not respond to second-line therapy；
* CD19 expression was positive by immunohistochemistry or flow cytometry (accept the results of this peripheral blood mononuclear cells or previous report from a Class A tertiary hospital before peripheral blood collection);
* If the subject has progressed or relapsed after prior CD19 CAR-T cell therapy, the planned apheresis phase should be at least 1 month after that, or the subject has been treated with other biologics, but is in the washout period;
* At least one measurable lesion at baseline, according to the Preliminary Assessment, staging and Response Assessment recommendations for Hodgkin's and non-Hodgkin's lymphoma (2014 edition);
* Expected survival time greater than 12 weeks;
* ECOG score 0-1 (subjects with central nervous system diseases caused by leukemia or lymphoma need to be determined by the investigator);
* Organ function：

  1. Complete blood count (CBC) test [the following criteria should be met within 24 hours prior to apheresis, and supportive treatment such as transfusion, platelet transfusion, cell growth factor (except recombinant erythropoietin) should be avoided within 7 days prior to detection]

     * Lymphocyte count ≥ 0.5×109/L (except for those receiving bridging chemotherapy);
     * Platelet count ≥ 25×109/L;
     * Hemoglobin ≥ 70.0 g/L
  2. Blood Biochemistry:

     * Serum creatinine (Scr) ≤ 1.5 x ULN, or
     * endogenous creatinine clearance ≥ 40 mL/min (using Cockcroft-Gault formula);
     * alanine aminotransferase (ALT) ≤ 2.5 x ULN;
     * aspartate aminotransferase (AST) ≤ 2.5 ×ULN;
     * Total bilirubin (TBIL) ≤ 2 ×ULN; Subjects with total bilirubin < 3 × ULN and direct bilirubin < 1.5× ULN with Gilbert-.Meulengracht syndrome could be included;
     * Serum lipase and amylase ≤ 1.5×ULN;
     * Alkaline phosphatase (ALP) ≤ 2.5 ×ULN;
     * In case of bone or liver metastasis, AST, ALT and ALP ≤ 5 ×ULN;
     * Prothrombin time (PT) extended ≤ 4 s, fibrinogen ≥ 1 g/L, activated partial thromboplastin time (APTT) ≤ 1.5 ×ULN;
  3. Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) > 91% in indoor air environment..
* Hemodynamic stability was determined by echocardiography or multichannel radionuclide angiography (MUGA) and LVEF ≥45％;
* Patients using the following drugs must meet the following conditions:

  1. Steroid: Therapeutic doses of steroids must be discontinued 2 weeks prior to Meta10-19 infusion. However, physiological replacement doses of steroids are permitted, hydrocortisone or its equivalent < 6-12mg/mm2/ day；
  2. Immunosuppressive agent: Any immunosuppressive drug must be stopped ≥4 weeks before the informed consent is signed;
  3. Stop all anti-proliferation therapies other than preconditioning chemotherapy in the 2 weeks before Meta10-19 infusion；
  4. Treatment for CNS disease must be stopped 1 week before Meta10-19 infusion (e.g., intrathecal methotrexate)
* The patient has recovered from the toxicity of the previous treatment, that is, the CTCAE toxicity grade is less than 1 (The exception is specific toxicity of grade 2 or less, such as hair loss, which the researchers have determined is not recoverable in a short period of time) is suitable for pretreatment chemotherapy and CAR-T cell therapy;
* Women of childbearing age and all male patients must consent to use a effective contraception for at least 12 months after Meta10-19 infusion and until two consecutive PCR tests show no more CAR T cells in vivo.

Exclusion Criteria:

* Patients with present or history of central nervous system diseases not associated with leukemia or lymphoma， such as seizures disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement;
* Patients who had received chemotherapy other than preconditioning chemotherapy within 2 weeks prior to Meta10-19 infusion;
* Patients who participated in other clinical trials within 30 days prior to enrollment;
* Patients with active hepatitis B (defined as hepatitis B surface antigen positive or hepatitis B core antibody positive, concomitant hepatitis B virus DNA level > 1000 copies/ml) or hepatitis C (HCV RNA positive);
* Patients with HIV antibody positive or treponema pallidum antibody positive;
* Patients with uncontrolled acute life-threatening bacterial, viral or fungal infections (e.g. positive blood cultures ≤72 hours before Meta10-19 infusion);
* History of unstable angina and/or myocardial infarction within 6 months prior to signing the informed consent; History of uncontrolled thrombotic events, major bleeding, or deep venous thrombosis (DVT) within 12 months prior to signing the informed consent;
* Patients with history of other malignancies, but the following conditions can be enrollment:

  1. Adequately treated basal or squamous cell carcinoma (requiring adequate wound healing before signing informed consent);
  2. Carcinoma in situ (DCIS) of cervical or breast cancer, which has been treated therapeutically, has shown no signs of recurrence for at least 3 years prior to the signing of the informed consent；
  3. The primary malignancy has been completely resected and in complete remission for ≥5 years；
* Women who are pregnant or breastfeeding (pregnancy tests for women of childbearing age are positive);
* History of QT interval prolongation or severe cardiac disease;
* Before signing the informed consent form, the ADA (FMC63) test was significantly positive (the test result was weakly positive, and it was necessary to discuss with the investigator whether to rule it out);
* Other conditions that the investigator considered should not be enrolled in this clinical study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
MTD | MTD will be determined based on DLTs observed during the first 35 days of study treatment.
  Determine the Maximal Tolerable Dose(MTD).
Objective response rate (ORR) | Within 3 months following infusion of Meta10-19.
  Measure Tumor response rate (including CR and PR).

SECONDARY OUTCOMES:
Concentration of CAR-T cells | Up to 12 months after CAR-T treatment.
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion.
Pharmacodynamics of CAR-T cells | Up to 28 days after infusion.
  Concentration levels of CAR-T related serum cytokines such as CRP, IL-6, INF-γ at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No